CLINICAL TRIAL: NCT03475914
Title: Characterization of Cutaneous Microbiota and Evaluation of the Antimicrobial Peptides Roles in the Psoriasis Etiopathogenesis
Brief Title: Characterization of Cutaneous Microbiota in the Psoriasis Pathogenesis
Acronym: MICROBIOTA
Status: Completed | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: MICROBIOTA
Record Dates: First submitted 2018-02-15; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-02

CONDITIONS: Psoriasis
Keywords: Psoriasis Guttate, Psoriasis vulgaris
MeSH Terms: conditions — Psoriasis; Guttate Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Biospecimen Retention: Samples With DNA — From each participant, a punch was used to obtain a cutaneous sample from both a lesioned and healthy skin area of 2 mm2 belonging t the left gluteus, for a total of 48 biological samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Psoriasis vulgaris: Pathological conditions stable for at least 1 month before collection. One punch biopsy from each patient, was taken from a big reddish and scaly plaque and another punch biopsy from the perilesional healthy skin.
- Psoriasis guttate: One punch biopsy from each patient, was taken from a small reddish and scaly plaque and another punch biopsy from the perilesional healthy skin.
- Healthy skin of psoriasis vulgaris: Healthy skin area of 2mm2 belonging to the left gluteus from patients affected by psoriasis vulgaris
- Healthy skin of psoriasis guttate: Healthy skin area of 2mm2 belonging to the left gluteus rom patients affected by psoriasis guttate

SUMMARY:
The skin harbors a complex and dynamic microbiota constituted by numerous microorganisms that live in symbiosis with the host. The specific etiology of psoriasis is still not-well understood; nonetheless several studies highlighted that that the skin microbiota could have a pivotal role in the maintenance and/or progression of the disease, acting as microbial predictor of psoriasis however.

The aim of the present study was to characterize the microbiota of cutaneous biopsies associated to guttate and vulgaris psoriasis, both considering lesion and healthy skin belonging to the same psoriatic subject.

DETAILED DESCRIPTION:
Twelve individuals with guttate psoriasis and 12 individuals with vulgaris psoriasis have been enrolled at Dermatological Unit of IRCCS Galeazzi Institute, Milan.

Patients selected for the psoriasis vulgaris group had a course of disease stable for at least 1 month before collection. The second group presented guttate psoriasis, defined as "eruptive", that is characterized by a rapid appearance and worsening of the clinical presentation within the month preceding the visit.

From each participant, a punch was used to obtain a cutaneous sample from both a lesion and healthy skin area of 2 mm2 belonging to the left gluteus, for a total of 48 biological samples. Participants were selected and included in the study according to the following criteria: i) over 18 years of age; ii) use of a free-preservatives soap with moisturizing function; iii) no use of probiotics; iv) no use of antibiotics; v) no treatment with corticosteroids, biological drugs, methotrexate or retinoids in the month prior the sampling; vi) no use of topical corticosteroids, vitamin D derivatives or phototherapy; vi) no chronic or systemic infections; vii) no cutaneous acute infections; viii) no allergy to pollen, food and drugs ix) no pets. Informed consent was obtained from all subjects.

A metagenomics approach, performed by the use of Ion torrent Personal machine, were used to investigate the bacterial composition of the skin microbiota associated to each samples collected.

After sequencing, the data analysis were focused on the bacterial biodiversity and microbial networks existing in the skin microbiota to evaluate a hypothetical role of bacteria in the complex pathophysiological mechanisms involved in psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age;
* use of a free-preservatives soap with moisturizing function, applied once a day;pets.

Exclusion Criteria:

* no use of probiotics in the month prior the sampling;
* no use of antibiotics in the month prior the sampling;
* no treatment with corticosteroids, biological drugs, methotrexate or retinoids in the month prior the sampling;
* no use of topical corticosteroids, vitamin D derivatives or phototherapy in the month prior the sampling;
* no chronic or systemic infections;
* no cutaneous acute infections during sampling;
* no allergy to pollen, food and drugs
* no pets.

Min Age: 18 Years | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Twelve individuals with guttate psoriasis and 12 individuals with vulgaris psoriasis have been enrolled at Dermatological Unit of IRCCS Galeazzi Institute, Milan.
  Patients selected for the psoriasis vulgaris group had a course of disease stable for at least 1 month before collection. The second group presented guttate psoriasis, defined as "eruptive", that is characterized by a rapid appearance and worsening of the clinical presentation within the month preceding the visit.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Psoriasis Area and Severity Index (PASI) | 1 year
  It is a measurement of psoriasis severity .

SECONDARY OUTCOMES:
Chao's index | 1 year
  It is a measure of bacterial biodiversity
Microbial abundance | 1 year
  It is a measure of bacterial amount
Spearman's correlation | 1 year
  It a measure of the bacterial interactions
Shannon's index | At the beginning of the study
  It is a measure of bacterial biodiversity
Simpson's index | 1 year
  It is a measure of bacterial biodiversity

IPD SHARING:
Plan to Share IPD: No